CLINICAL TRIAL: NCT03370562
Title: Dexmedetomidine After Cesarean for the Treatment of Nausea and Shivering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Hess, Staff Anesthesiologist, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017P000517
Record Dates: First submitted 2017-11-27; First posted 2017-12-12 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Shivering; Nausea and Vomiting, Postoperative
Keywords: dexmedetomidine; cesarean; spinal anesthesia
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study medication provided in blinded syringe labeled with study number
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Patient will receive 10 mcg of dexmedetomidine in 5 ml of normal saline, administered by slow intravenous injection
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Patient will receive 5 ml of normal saline, administered by slow intravenous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Administration of 10 mcg intravenous dexmedetomidine
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Placebo — Administration of normal saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This is a randomized double blinded trial to determine if a small dose of dexmedetomidine can prevent and relieve nausea and shivering, two of the more common complaints after cesarean delivery.

DETAILED DESCRIPTION:
This study is a randomized, placebo controlled, double blind evaluation of the use of a single dose of dexmedetomidine for the prevention of shivering and nausea after cesarean delivery. It is hypothesized that patients who receive dexmedetomidine (as compared to placebo) will have a reduced severity of postoperative shivering and nausea.

Study subjects will be have a scheduled cesarean section. They will receive written, informed consent obtained before surgery. After enrollment, patients will receive spinal anesthesia consisting of 11.25mg bupivacaine, 25 mcg of fentanyl, and 250 mcg of morphine. All IV fluid will be warmed.

After delivery of the neonate, delivery of the placenta, and assurance of adequate uterine tone, patients will be randomized in a 1:1 fashion to receive a blinded study syringe consisting of either placebo saline, or 10 mcg of dexmedetomidine.

Study outcomes will be measured on an 11-point Likert scale assessing shivering, nausea, pain, pruritus, and sedation. Assessments will be performed on admission to the recovery room, and at 30 and 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean delivery
* ≥ 18 years of age
* Singleton pregnancy
* Term delivery (37 weeks or greater gestation)
* Spinal or combined spinal-epidural anesthesia is planned

Exclusion Criteria:

* Non-elective cesarean delivery
* Receiving misoprostil or carboprost
* Postpartum hemorrhage greater that 1000cc
* Chronic opioid use
* History of chronic nausea or itching in pregnancy
* Receiving medications for nausea
* Inability to provide written informed consent
* Receiving of any of the following medications intraoperatively: misoprostil, carboprost, medications for nausea
* Postpartum hemorrhage greater that 1000cc

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females will be enrolled
Enrollment: 100 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Shivering measured by Visual analogue score | 60 minutes
  Severity of patient shivering measured on a 10-centimeter line with 0 cm representing none and 10 cm representing worst possible
Postoperative nausea and vomiting measured by Visual analogue score | 60 minutes
  Severity of postoperative nausea and vomiting measured on a 10-centimeter line with 0 cm representing none and 10 cm representing worst possible

SECONDARY OUTCOMES:
Pain measured by Visual analogue score | 60 minutes
  Severity of incisional pain measured on a 10-centimeter line with 0 cm representing none and 10 cm representing worst possible
Pruritus measured by Visual analogue score | 60 minutes
  Severity of postoperative pruritus measured on a 10-centimeter line with 0 cm representing none and 10 cm representing worst possible
Sedation measured by Visual analogue score | 60 minutes
  Severity of postoperative sedation measured on a 10-centimeter line with 0 cm representing none and 10 cm representing worst possible
Dry mouth measured by Visual analogue score | 60 minutes
  Severity of patient complaint of dry mouth measured on a 10-centimeter line with 0 cm representing none and 10 cm representing worst possible

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Hess, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No